CLINICAL TRIAL: NCT07174804
Title: Investigating the Role of Yoga in Alleviating Chromosomal Translocations in Security Guards of Chandigarh Police Who Are Responsible for the Safety of VIPs
Brief Title: Chromosomal Translocations in Chandigarh Police
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Swami Vivekananda Yoga Anusandhana Samsthana (Unknown)
Responsible Party: Principal Investigator, Sheetal Sharma, Principal Investigator, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IEC-08/2019-1290
Record Dates: First submitted 2025-09-03; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Chromosomal Translocations
MeSH Terms: conditions — Translocation, Genetic | interventions — Yoga; Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IAYT Group (Yoga Group) (Experimental): This group will be formed from highly stressed individuals and will follow yoga protocol as intervention for three months.
  Interventions: Other: Yoga (IAYT) Intervention
- Control Group (No Intervention): This group will be formed from highly stressed individuals and will not follow yoga protocol as intervention.

INTERVENTIONS:
Other: Yoga (IAYT) Intervention — Yoga practice for a period of three months
  Arms: IAYT Group (Yoga Group)

SUMMARY:
The goal of this Non-Randomized Control Trial is to evaluate the prevalence of chromosomal translocations in occupationally stressed subjects and the molecular impact of yoga on such translocations and DNA damage response and repair in security guards of Chandigarh Police. The main questions it aims to answer are:

Does yoga has any role in alleviating chromosomal translocations in healthy but occupationally stressed subjects? Does practice of yoga has any impact on molecular markers related to DNA damage response and repair before and after Yoga intervention in highly stressed individuals? Researchers will compare Control Group and Yoga group before and after Yoga intervention.

Participants will be divided into two groups Control Group and Yoga Group. Yoga Group will be given yoga intervention for 3 months, 5 days a week and for 65 minutes in a day. Control Group will follow their daily routine without following the intervention. Before and after the intervention, blood samples will be collected from the participants of both groups and analysed for chromosomal translocations and DDRR markers.

DETAILED DESCRIPTION:
Definition of the problem: Evaluate the molecular impact of yoga on DNA damage response and repair on security guards of Chandigarh Police

Objectives:

1. Analysis of molecular markers related to DNA damage response and repair before and after the practice of yoga on Chandigarh Police
2. To examine the molecular mechanism by which yoga may modulate DNA damage response and repair.

Recruitment of individuals: Department of Police, Chandigarh has agreed to help the investigators on this aspect. Policemen working for Chandigarh Police will be chosen based on the inclusion and exclusion criteria.

Subjects: Those security guards (age: >20 and <60) who are willing to consent to participate in this study will be screened for moderate and higher stress on Cohen's PSS, according to inclusion criteria and randomly divided between Intervention (Yoga Group) and Control Group.

Sample Size: The sample size of 206 was calculated for 99% confidence level (reliability coefficient = 2.58), at the alpha level of 0.05, a power of 0.95, and a relative precision of 0.2, derived from a pilot study done on breast cancer patients and yoga practitioners (Ram et al, 2013). Assuming a 10% drop out rate, a total of 229 subjects will be recruited.

Design of the study In a randomized control trial (RCT), participants are allocated randomly between intervention and control groups to compare the treatments, which enables statistical control over the influences imparted by the aforementioned treatments. In the present study, the policemen who satisfy the study's eligibility criteria and willing to consent to participate in this study will be enrolled, grouped randomly in intervention and control groups, and assessed for the dependent variables of the study before and after the Integrated Yoga intervention period.

Variables Socio-demographic details - age, diet, alcohol consumption, etc. Evaluation of stress level on Cohen's Perceived Stress Scale (pre and post intervention) (Cohen, Kamarck & Mermelstein, 1983) Evaluation of stress level using vital parameters: Blood pressure and resting heart rate of participants will be recorded pre and post intervention.

Evaluation of stress level using molecular parameters: (pre and post intervention) 10 ml of blood will be withdrawn from the subjects by trained phlebotomists, and coded. WBCs and plasma will be separated using standard protocols and stored at -80℃. Plasma will be utilized to assess the levels of cortisol.

Assessment of chromosomal translocations: (pre and post intervention) Genomic DNA will be extracted from WBCs isolated, and tested for chromosomal translocations using PCR assay. Isolated genomic DNA will be subjected to nested PCR using primers specifically designed to check for t(14;18) and t(11;14) translocations.

Assessment of DDR and DNA repair:

Immunofluorescence: Isolated PBMCs will be subjected to DDR analysis by immunofluorescence. For this, these cells will be fixed and stained with various DDR markers like γH2AX, 53BP1, pATM.

Gene expression analysis: Total RNA will be isolated from these cells; cDNA will be synthesized and the expression of following DDR and DNA repair genes will be performed using real-time PCR: RAD51, MRE11, RAD50, NBS1, KU70, LIGASE IV, PARP1 Comet assay: Cells will be used to perform both the neutral as well as alkaline comet assay to assess for the number of single- and double-strand breaks.

Telomeric length: Relative telomere length (TL) using quantitative polymerase chain reaction (qPCR) will be performed on genomic DNA isolated from control and group blood samples and will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Individuals scoring more than 15 points on Cohen's scale. Once these subjects' consent to enrol, each one of them will be coded to maintain anonymity.

Exclusion Criteria:

* Individuals with complications in co-morbid conditions like Diabetes, Cirrhosis, etc.
* Individuals of age less than 25 or more than 60 years.
* Individuals who do not consent to be a part of this study.
* Individuals who fail to comply with the yoga protocol in Intervention Group.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 203 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of t(14;18) translocations using Nested PCR method | 3 months
  Both control and yoga group will be assessed for prevalence of chromosomal translocations t(14;18) before and after yoga (IAYT) intervention. This prevalence will be measured as relative band intensity for each individual and will be compared for before and after IAYT intervention, and also for between the groups after intervention.

SECONDARY OUTCOMES:
Cohen's Perceived Stress Scale | 3 months
  Both groups will be assessed for perceived stress before and after yoga (IAYT) intervention.
Six Letter Cancellation Test (SLCT) | 3 months
  Both groups will be assessed for SLCT scores to measure neuropsychological performance before and after yoga (IAYT) intervention
Trail Making Test (TMT) | 3 months
  Both groups will be assessed for TMT time to measure neuropsychological performance before and after yoga (IAYT) intervention
Serum cortisol level using enzyme-linked immunosorbent assay | 3 months
  Both groups will be assessed for serum cortisol levels before and after yoga (IAYT) intervention. This will be measured with the help of standard curve in ng/mL for each individual and will be compared for before and after IAYT intervention, and also for between the groups after intervention.
Relative Telomere Length using Real-Time PCR | 3 months
  Participants will be assessed for Relative Telomere Length before and after yoga (IAYT) intervention. This will be measured in fold change using qPCR for each individual.

CONTACTS AND LOCATIONS:
Overall Officials: Sheetal Sharma, Principal Investigator — Postgraduate Institute of Medical Education & Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Yes
Age, Occupation, Gender, Neuropsychological Data, Cortisol levels, Relative Telomere Length and chromosomal Translocations
Supporting Information: Study Protocol, SAP, ICF
Time Frame: September 2026 to December 2026
Access Criteria: Access to individual participant data will be granted to qualified researchers affiliated with academic or non-profit institutions. Requests must include a research proposal describing the purpose of use. Requests will be reviewed by the principal investigator and must comply with local and international data protection regulations. Data will be shared under a data use agreement to ensure confidentiality and non-commercial use.

DOCUMENTS (3):
  • Study Protocol (2020-02-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT07174804/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT07174804/SAP_001.pdf
  • Informed Consent Form (2020-02-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT07174804/ICF_002.pdf